CLINICAL TRIAL: NCT07175012
Title: ELECTROVEST: Electro-Stimulation Vibratory Vest for Pulmonary Rehabilitation in Patients With Chronic Respiratory Diseases
Acronym: Electrovest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Rafael Rivilla Rivilla, Physiotherapist - Clinical Researcher, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EXP - 00111621 / ITC-20181118
Record Dates: First submitted 2025-07-14; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Cystic Fibrosis (CF); Bronchiectasis Adult; Asthma Bronchiale
Keywords: Electrostimulation; High-Frequency Chest Wall Oscillation (HFCW; Airway Clearance; Chronic Respiratory Diseas; Respiratory Physiotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, two-period crossover trial. Each participant will undergo two treatment phases: one with the investigational device (ELECTROVEST) and one with the standard HFCWO vest (The Vest®). A 30-day washout period will separate the two phases. Each participant will serve as their own control, allowing for intra-individual comparisons of outcomes such as sputum production, pulmonary function, respiratory muscle strength, and tolerability.
Masking Description: This is an open-label study. No masking was applied to participants, care providers, investigators, or outcome assessors due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELECTROVEST Intervention (Experimental): Participants in this arm will receive airway clearance therapy using the ELECTROVEST, a wearable device that combines high-frequency chest wall oscillation (HFCWO) with surface neuromuscular electrostimulation (EEM). The intervention will be administered alongside standard fluid and aerosol therapy. This phase is designed to evaluate the device's safety, effectiveness, and tolerability.
  Interventions: Device: ELECTROVEST
- Standard HFCWO Therapy (Control) (Active Comparator): Participants in this arm will receive standard airway clearance therapy using a high-frequency chest wall oscillation (HFCWO) vest device, either The Vest® Model 105 or the AffloVest®. The therapy will be combined with fluid and aerosol therapy and will serve as the comparator for evaluating the ELECTROVEST intervention. Participants will undergo this treatment after a 30-day washout period.
  Interventions: Device: The Vest® Model 105

INTERVENTIONS:
Device: ELECTROVEST — A wearable vest device that delivers airway clearance therapy through high-frequency chest wall oscillation (HFCWO) combined with surface neuromuscular electrostimulation (EEM). The session includes a 2-minute warm-up phase at 4 Hz, 16 minutes of active stimulation at 8 Hz, and a 2-minute recovery phase at 4 Hz (total duration: 20 minutes). The intervention is administered during supervised physiotherapy sessions to promote mucociliary clearance and respiratory muscle activation in patients with chronic respiratory diseases.
  Other Names: Electrostimulation Vibratory Vest
  Arms: ELECTROVEST Intervention
Device: The Vest® Model 105 — A conventional airway clearance therapy using a commercial high-frequency chest wall oscillation (HFCWO) device (The Vest® Model 105 or AffloVest®). The session includes a 2-minute warm-up phase at 13 Hz, 16 minutes of treatment at 20 Hz, and a 2-minute cool-down at 13 Hz (total duration: 20 minutes). This intervention serves as the active comparator in the crossover trial.
  Other Names: Standard HFCWO Therapy
  Arms: Standard HFCWO Therapy (Control)

SUMMARY:
This study will evaluate the effectiveness, safety, and tolerability of a novel wearable device, the ELECTROVEST, designed to improve airway clearance in patients with chronic respiratory diseases. The ELECTROVEST will integrate high-frequency chest wall oscillation (HFCWO) with surface neuromuscular electrostimulation. This crossover clinical trial will compare the performance of the ELECTROVEST with a standard HFCWO vest (The Vest®) in adult patients. Primary outcomes will include sputum expectoration and patient-reported comfort. The study will aim to determine whether this new system can optimize bronchial hygiene.

DETAILED DESCRIPTION:
This is a prospective, crossover pilot study designed to evaluate the safety, efficacy, and tolerability of a novel respiratory therapy device, ELECTROVEST, in adult patients diagnosed with chronic respiratory diseases featuring bronchial hypersecretion, such as COPD, bronchiectasis, cystic fibrosis, and asthma.

ELECTROVEST is a wearable vest that integrates high-frequency chest wall oscillation (HFCWO) with surface neuromuscular electrical stimulation (NMES). This dual-action therapy aims to enhance airway clearance while also stimulating respiratory musculature.

The study will enroll 20 patients, using a non-probabilistic, intentional sampling strategy. Each participant will undergo two intervention phases, acting as their own control. The phases are separated by a 30-day washout period to minimize carryover effects.

Phase 1 (ELECTROVEST intervention): Participants receive standard fluid and aerosol therapy followed by vibratory therapy delivered by the ELECTROVEST device. Sessions include:

Warm-up phase: 2 minutes at 4 Hz

Active treatment: 16 minutes at 8 Hz

Cool-down phase: 2 minutes at 4 Hz

Phase 2 (Control intervention): Participants receive the same fluid and aerosol therapy, followed by vibratory therapy using standard HFCWO systems (The Vest® Model 105 ). The session follows:

Warm-up: 2 minutes at 13 Hz

Active treatment: 16 minutes at 20 Hz

Cool-down: 2 minutes at 13 Hz

Both interventions are conducted under clinical supervision. The effects will be assessed through pulmonary function tests, respiratory muscle strength, sputum analysis, oxygenation and hemodynamics, patient-reported symptoms, and blood biomarkers.

Pulmonary function and muscle strength will be measured before and 10 minutes after each intervention (FEV₁, DLCO, PImax, PEmax, SNIP). Sputum production and quality will be assessed by weight and purulence (Murray scale). Exercise tolerance will be evaluated via the 6-minute walk test.

Blood markers will be obtained before and 48 hours after each intervention, including:

Creatine phosphokinase (CPK-MM, CPK-BB)

C-reactive protein (CRP)

Peripheral leukocyte count

Creatinine, urea, albumin

Estimated glomerular filtration rate (eGFR)

Venous lactate

Monitoring during sessions includes:

Oxygen saturation (SpO₂)

Heart rate

Discomfort and dyspnea assessed via a visual analogue scale (VAS, 0-10), recorded at baseline, 5 minutes, and post-treatment.

This trial aims to identify physiological responses, tolerability, and short-term safety signals, while generating preliminary data on the potential dual utility of the ELECTROVEST device as a mucociliary clearance and respiratory muscle stimulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Respiratory Diseases Diagnosed with chronic respiratory disease with bronchial hypersecretion: COPD, cystic fibrosis, bronchiectasis, or asthma
* Age >16 years
* Clinically stable (no exacerbations in past 4 weeks)

Exclusion Criteria:

* Risk of pneumothorax and/or barotrauma
* Risk or history of hemoptysis
* On active waiting list for lung transplant or surgery
* Musculoskeletal or other limiting condition
* Diagnosis of osteoporosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Volume of Expectorated Sputum | Immediately post-intervention (within 1 hour)
  Total sputum weight (in grams) collected during and within 1 hour after each airway clearance session
Discomfort Level (VAS Score) | Immediately after each intervention session
  Subjective discomfort assessed using a 0-10 visual analogue scale (VAS), where 0 indicates no discomfort and 10 indicates maximum discomfort.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 Second (FEV1) | Baseline and 24-48 hours after each intervention.
  FEV1 measured via spirometry, according to ATS/ERS standards.
Maximal Inspiratory Pressure (PImax) | Baseline and 24-48 hours after each intervention.
  Respiratory muscle strength measured in cmH2O using MicroRPM (Carefusion)
Maximal Expiratory Pressure (PEmax) | Baseline and 24-48 hours after each intervention.
  Respiratory muscle strength measured in cmH2O using MicroRPM (Carefusion)
Six-Minute Walk Distance (6MWD) | Baseline and 24-48 hours after each intervention.
  Distance walked in meters during the 6-minute walk test as a measure of functional capacity.
DLCO (Diffusing Capacity for Carbon Monoxide) | Baseline and 24-48 hours after each intervention.
  Measured using single-breath technique, following ATS/ERS 2017 guidelines.
Inflammatory and Muscle Biomarkers | Baseline and 24-48 hours after each intervention.
  Blood markers including creatine phosphokinase (CPK) and C-reactive protein (CRP), measured through standard blood analysis.
Maximal Nasal Inspiratory Pressure (SNIP) | Baseline and 24-48 hours after each intervention.
  Nasal inspiratory pressure assessed using the SNIP test (Sniff Nasal Inspiratory Pressure) to evaluate inspiratory muscle strength. Unit measure cmH₂O.
Estimated Glomerular Filtration Rate (eGFR) | Baseline and 24-48 hours after each intervention.
  Renal function assessed using estimated glomerular filtration rate (eGFR), calculated using the Cockcroft-Gault formula based on blood creatinine, age, weight, and sex.
Health-Related Quality of Life (CASA-Q) | Baseline and 24-48 hours after each intervention.
  Health status and cough-related quality of life evaluated using the CASA-Q questionnaire (Cough and Sputum Assessment Questionnaire). Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided whether individual participant data (IPD) will be shared. The study team is currently evaluating the feasibility of anonymizing and storing IPD in a secure repository in accordance with institutional and ethical guidelines.

REFERENCES:
- [Derived] Rivilla Rivilla R, Mendez Alonso AY, Roque Betancourt E, Vazquez Sanchez RM, Ortiz Molina I, Bonail Acuna B, Elena Perez MDM, Tejero Garcia S, Diaz Gutierrez F, Quintana Gallego E, Giraldez Sanchez MA, Cejudo Ramos P. Electrovest(R): A novel portable electro-vibratory device for airway clearance in chronic hypersecretory lung diseases. Pulmonology. 2025 Dec 31;31(1):2594888. doi: 10.1080/25310429.2025.2594888. Epub 2025 Dec 1. PMID 41324124